CLINICAL TRIAL: NCT03499132
Title: Influence of Different Anesthetic Procedures on Sleep Disorder Breathing in Adult Patients Undergoing Elective Surgery
Brief Title: Influence of Different Anesthetic Procedures on Sleep Disorder Breathing
Status: Completed | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, M.D., Ph.D., St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: IIT/2017/30
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: anesthesia, obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- General anesthesia (with opioids): orthopedic surgery plus general anesthesia
  Interventions: Procedure: anesthesia
- Epidural anesthesia (without opioids): orthopedic surgery plus epidural anesthesia (without opioids use)
  Interventions: Procedure: anesthesia
- Subarachnoid anesthesia (with opioids): orthopedic surgery plus subarachnoid anesthesia (plus intrathecal opioid)
  Interventions: Procedure: anesthesia
- Regional anesthesia (without opioids): orthopedic surgery plus regional anesthesia (peripheral nerve block, continous or single shot, without opioid use)
  Interventions: Procedure: anesthesia

INTERVENTIONS:
Procedure: anesthesia — Different anesthetic procedures

SUMMARY:
Obstructive sleep apnea (OSA) is a common form of sleep disordered breathing characterized by partial or complete upper airway obstructions during sleep. OSA is associated with major comorbidities and perioperative complications. These complications are caused not only by the OSA itself, but also by exacerbations of this syndrome during the perioperative period (1). Benzodiazepines, volatile anesthetics and opioids may lead to lower hypoxia and hypercapnia sensitivity and may cause respiratory depression (2-5). Therefore, preference of neuraxial blockades and avoidance of opioids has been suggested for patients with OSA (6). However, there is still lack of evidence to evaluate the effects of various anesthesia procedures on OSA (6,7). We hypothesize different anesthetic procedures will have different effect on OSA exacerbations in the postoperative period. Accordingly, the aim of this study is to compare the number of sleep disordered breathing episodes in the postoperative period in patients with different anesthetic procedures.

ELIGIBILITY:
Inclusion Criteria:

* elective orthopedic surgery

Exclusion Criteria:

* already diagnosed sleep disorder breathing
* continuous positive airway pressure therapy
* tracheostomy
* American Society of Anesthesiologists class IV-V

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing elective orthopedic surgery
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index change | 4 nights after surgery
  Changes (post-pre) in apnea-hypopnea index 4 nights post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cundrle, M.D., Ph.D., Principal Investigator — St. Anne's University Hospital Brno
Locations (1):
- St. Anne's University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung F, Liao P, Elsaid H, Shapiro CM, Kang W. Factors associated with postoperative exacerbation of sleep-disordered breathing. Anesthesiology. 2014 Feb;120(2):299-311. doi: 10.1097/ALN.0000000000000041. PMID 24158050
- [Background] Alexander CM, Gross JB. Sedative doses of midazolam depress hypoxic ventilatory responses in humans. Anesth Analg. 1988 Apr;67(4):377-82. PMID 3354874
- [Background] Weil JV, McCullough RE, Kline JS, Sodal IE. Diminished ventilatory response to hypoxia and hypercapnia after morphine in normal man. N Engl J Med. 1975 May 22;292(21):1103-6. doi: 10.1056/NEJM197505222922106. PMID 1128555
- [Background] Dahan A, van den Elsen MJ, Berkenbosch A, DeGoede J, Olievier IC, van Kleef JW, Bovill JG. Effects of subanesthetic halothane on the ventilatory responses to hypercapnia and acute hypoxia in healthy volunteers. Anesthesiology. 1994 Apr;80(4):727-38. doi: 10.1097/00000542-199404000-00004. PMID 8024126
- [Background] van den Elsen M, Dahan A, DeGoede J, Berkenbosch A, van Kleef J. Influences of subanesthetic isoflurane on ventilatory control in humans. Anesthesiology. 1995 Sep;83(3):478-90. doi: 10.1097/00000542-199509000-00006. PMID 7661348
- [Background] American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):268-86. doi: 10.1097/ALN.0000000000000053. No abstract available. PMID 24346178
- [Background] Roesslein M, Chung F. Obstructive sleep apnoea in adults: peri-operative considerations: A narrative review. Eur J Anaesthesiol. 2018 Apr;35(4):245-255. doi: 10.1097/EJA.0000000000000765. PMID 29300271